CLINICAL TRIAL: NCT00008502
Title: Genetic Analysis of Familial Keloids
Status: Completed | Type: Observational
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 010062; 01-DK-0062
Record Dates: First submitted 2001-01-12; First posted 2001-01-15 (Estimated); Last update posted 2021-08-27 (Actual); Status verified 2021-08

CONDITIONS: Keloid
Keywords: Genetics; African Americans; Skin; Keloids
MeSH Terms: conditions — Keloid

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Cross-Sectional

GROUPS / COHORTS (3):
- 18 years of age or older: without keloids
- family members over 12 years of age: who have either classic or non-classic keloids
- Probands: original participants who have had a classic (butterfly-shaped or wound-overflowing) keloidfor at least one year

SUMMARY:
The purpose of this study is to identify the gene or genes responsible for keloid formation. Keloids are raised scars on the skin that form after a minor injury. A tendency to develop keloids often runs in families, suggesting a possible genetic basis.

People who have had a classic (butterfly-shaped or wound-overflowing) keloid for at least one year may be eligible for this study. In addition to these probands (original participants), family members over 12 years of age who have either classic or non-classic keloids and those 18 years of age or older without keloids may participate.

Probands and family members with keloids will have a medical history focusing on skin problems-particularly keloids-and a skin examination. In some cases, with the subject s permission, photos of the keloids will be taken. All participants will have 35 milliliters (about 2 tablespoons) of blood drawn for DNA (genetic) testing and for measurement of blood proteins, including cytokines, which can affect other tissues and cause scarring. Part of the blood sample will be used for additional genetic studies unrelated to keloids. The samples will be coded for confidentiality.

DETAILED DESCRIPTION:
Keloids represent a pathologic fibrosis which occurs in the skin after trauma and which grow beyond the boundaries of injury. Keloids occur in people of all racial backgrounds; however, individuals of African descent are more susceptible to the disease. A familial disposition to keloid formation has long been recognized, but the genetic basis for this racial and familial predisposition has not been identified. We hypothesize that the increased risk is a direct result of one or more disease susceptibility genes. We will pursue two approaches, which are presented as two study modules. In module 1, we will carry out a family study. We will identify affected pedigrees, each containing at least 3 individuals with keloids. Blood will be obtained and Epstein Barr virus-transformed permanent B cell lines will be established. We anticipate taking two analytic strategies. We will use candidate gene analysis, focusing initially on the CBP and TGF1B genes and a recently identified locus on chromosome 14, and we will use genome-wide markers to identify possible disease gene loci. In module 2, we will perform a genome scan to address the hypothesis that one or more African origin genetic variants account for the excess prevalence of keloids among African Americans. We will carry out a mapping by admixture linkage disequilibrium (MALD) scan, in order to find genetic regions where differences in the distribution of particular tagging single nucleotide polymorphisms (SNPs) between keloid cases and controls indicate excess African ancestry. Further analysis of these loci will be carried out to identify the causative genetic variants.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Proband: must have a butterfly-shaped or wound-overflowing keloid, present for at least one year (this description represents classic keloid, and avoids hypertrophic scar)
  2. Affected family members: all family members of the proband who have either classic keloids, as described above, or non-classic keloids, such as ball shaped-keloids on the ear.
  3. Unaffected family members: all family members who lack keloids.
  4. Impaired subjects for whom a legal guardian provides consent.
  5. Pregnant women.

EXCLSUION CIRTERIA:

1. Subjects who are unwilling or unable to give informed consent or assent.
2. Impaired individuals from whom it not possible to obtained parental consent (minors) or guardian consent (adults).
3. Keloid patients who have <3 relatives with keoids.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: People who have had a classic (butterfly-shaped or wound-overflowing) keloid for at least one year may be eligible for this study. In addition to these probands (original participants), family members over 12 years of age who have either classic or non-classic keloids and those 18 years of age or older without keloids may participate.
Sampling Method: Non-Probability Sample
Enrollment: 106 (Actual)
Dates: Start 2001-08-14 (Actual); Primary Completion 2017-11-28 (Actual); Study Completion 2017-11-28 (Actual)

PRIMARY OUTCOMES:
Finding a genetic locus | 12/01/2018
  The purpose of this study is to identify the gene or genes responsible for keloid formation

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey B Kopp, M.D., Principal Investigator — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2001-DK-0062.html